CLINICAL TRIAL: NCT01310322
Title: An Open, Partly Randomised, Four-way Cross-over Study in Healthy Subjects and in Patients With Mild Allergic Asthma to Investigate the Bioavailability and Basic Pharmacokinetics of a Single Dose of AZD5423 When Administered Intravenously, Orally, Inhaled Via SPIRA Nebuliser or Inhaled Via I-neb® AAD Systems
Brief Title: A Study in Healthy Subjects and Mild Asthmatics to Investigate Pharmacokinetics of AZD5423 When Administered in Different Ways
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D2340C00008
Record Dates: First submitted 2011-02-17; First posted 2011-03-08 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy; Asthma
Keywords: Phase I; Healthy male volunteers; mild asthmatics; pharmacokinetics; Bioavailability and AUC; Level of AZD5423 in your blood
MeSH Terms: conditions — Asthma | interventions — 2,2,2-trifluoro-N-(1-((1-(4-fluorophenyl)-1H-indazol-5-yl)oxy)-1-(3-methoxyphenyl)-2-propanyl)acetamide

ARMS (4):
- 1 (Experimental): AZD5423 iv
  Interventions: Drug: AZD5423
- 2 (Experimental): AZD5423 inhalation, Spira
  Interventions: Drug: AZD5423
- 3 (Experimental): AZD5423 inhalation I-neb
  Interventions: Drug: AZD5423
- 4 (Experimental): AZD5423 oral
  Interventions: Drug: AZD5423

INTERVENTIONS:
Drug: AZD5423 — solution for injection, administered as intravenous infusion Corr to total dose of 250µg AZD5423
  Arms: 1
Drug: AZD5423 — nebuliser suspension, inhaled via Spira, corr to approximately 300 µg lung deposited dose AZD5423
  Arms: 2
Drug: AZD5423 — nebuliser suspension, inhaled via I-neb, corr to approximately 300 µg lung deposited dose AZD5423
  Arms: 3
Drug: AZD5423 — nebuliser suspension to be administered orally, corr to a total dose of 1200 µg AZD5423
  Arms: 4

SUMMARY:
A study in healthy subjects and mild asthmatics to investigate Pharmacokinetics of AZD5423 when administered in different ways.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy subjects and male asthma patients aged 18 to 45 years (inclusive)
* Have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive and rounding allowed) and weight between 50 and 100 kg (inclusive)
* Be able to inhale from the SPIRA nebuliser and I-neb® according to the provided instructions
* Asthma patients should fulfil the following criteria: Pre-bronchodilator forced expiratory volume at 1 second (FEV1) ≥70% of predicted normal value
* Asthma diagnosis according to GINA guidelines with a history of episodic wheeze and shortness of breath

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Any clinically relevant abnormal findings
* Current smokers
* Asthma patients: Worsening of asthma or respiratory infection within 6 weeks before screening
* Asthma patients: Use of inhaled, nasal, oral, rectal or parenteral corticosteroids within 30 days before first administration of investigational product and during the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD5423 measured by: Absolute bioavailability (F) | Pharmacokinetic (PK) sampling will be performed day 1 to day 5 for each treatment period
Pharmacokinetics of AZD5423 measured by: Pulmonary bioavailability (Fpulmonary) | Pharmacokinetic (PK) sampling will be performed day 1 to day 5 for each treatment period
Pharmacokinetics of AZD5423 measured by: Oral bioavailability after inhaled treatments (Foral) | Pharmacokinetic (PK) sampling will be performed day 1 to day 5 for each treatment period
Pharmacokinetics of AZD5423 measured by: Area under the plasma concentration-time curve from time zero to infinity (AUC). | Pharmacokinetic (PK) sampling will be performed day 1 to day 5 for each treatment period

SECONDARY OUTCOMES:
To compare the pharmacokinetics between healthy subjects and asthma patients and estimate the basic pharmacokinetic parameters of AZD5423 by measuring e.g. maximum plasma concentration, Cmax | Pharmacokinetic (PK) sampling will be performed day 1 to day 5 for each treatment period
To evaluate the safety and tolerability of AZD5423 measured by adverse events, laboratory variables, physical examination, electrocardiograms, blood pressure and pulse, and spirometry. | From screening to follow-up
  To evaluate the safety and tolerability of AZD5423 measured by (Adverse events) (Laboratory variables) (Physical examination) (Electrocardiograms) (blood pressure and pulse) (Spirometry)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, Dr, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Research Unit, London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1257&filename=D2340C00008.pdf